CLINICAL TRIAL: NCT03839654
Title: The Role and Mechanisms of Loop Gain and Associated Parameters in the Reversion of OSA Treated by Either CPAP or Cardiac Valve Replacement
Brief Title: Loop Gain in the Reversion of OSA Treated by Either CPAP or Cardiac Valve Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ning Ding, Principal Investigator, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2019-SR-016
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Obstructive Sleep Apnea of Adult; Heart Valve Diseases
Keywords: Obstructive Sleep Apnea; heart valve replacement; CPAP treatment; loop gain
MeSH Terms: conditions — Heart Valve Diseases; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: A total of 300 patients with rheumatic valvular heart disease waiting for cardiac valve replacement were screened for obstructive sleep apnea (OSA). Of them, 40 OSA patients were enrolled and randomly received CPAP treatment and non-CPAP treatment (20:20 patients). The CPAP treatment group received both baseline medicine and CPAP treatment for 7 days preoperatively. The non-CPAP treatment group only received baseline medicine treatment.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continuous positive airway pressure (Experimental): The CPAP treatment group received both baseline medicine and CPAP treatment for 7 days preoperatively.
  Interventions: Device: continuous positive airway pressure
- non-continuous positive airway pressure (No Intervention): The non-CPAP treatment group received baseline medicine treatment without CPAP treatment.

INTERVENTIONS:
Device: continuous positive airway pressure — The CPAP treatment group received both baseline medicine and CPAP treatment for 7 days preoperatively.
  Arms: continuous positive airway pressure

SUMMARY:
Sleep apnea including obstructive sleep apnea (OSA) and central sleep apnea (CSA), are common in patients with cardiovascular disease. The prevalence of OSA is 2%-4% in general population and 16%-47% in surgical-heart failure patients.

The previous studies found that the sleep apnea types shifted from OSA to CSA after continuous positive airway pressure (CPAP) treatment or from CSA to OSA after heart surgery (cardiac valve replacement/ repair or heart transplantation) without the mechanism illuminated clearly. The recent studies found that the loop gain (LG) could predict the effect of upper airway surgery and CPAP treatment on the reversion of OSA. However, in patients with valvular heart disease, whether LG and related parameters can predict the therapeutic efficacy of CPAP or cardiac valve replacement is not expounded clearly.

The investigators' previous study found that there were different outcomes of sleep apnea after cardiac valve replacement: elimination or consistent. But the corresponding non-anatomic mechanisms was not clear. The investigators' preliminary experiment showed that the LG and related parameters were not improved while OSA improved by CPAP treatment; however, the recovery of OSA after cardiac valve replacement was closed related to the improvement of LG and related parameters.

The investigators speculated that, 1. LG and related parameters could predict OSA outcome of CPAP treatment or cardiac valve replacement. 2. non-anatomic mechanisms including LG and associated parameters, contributed to CPAP treatment and cardiac valve replacement were different. In this study, the investigators aimed to explore the relationship between LG and, outcomes of OSA and the regarding non-anatomic mechanisms in patient with heart valve disease.

DETAILED DESCRIPTION:
Between January 31, 2020 and June 30, 2023, 300 patients with valvular heart disease waiting for cardiac valve replacement in Department of Cardiovascular Surgery were screened for obstructive sleep apnea (OSA) by full-night polysomnography. Of them, 40 OSA patients were enrolled and randomly received CPAP treatment and non-CPAP treatment (20:20).

The CPAP treatment group received both baseline medicine and CPAP treatment. The full-night CPAP treatment was conducted from 21:00 pm to 6:00 am for 7 days preoperatively. The non-CPAP treatment group received baseline medicine treatment. LG and related parameters were collected at the first day of treatment in non-CPAP group and both first and last day of treatment in CPAP group.

Sleep parameters including apnea-hypopnea index (AHI), mean and lowest SPO2, and clinical evaluations including New York Heart Association (NYHA) classes, electrocardiographic, echocardiographic, arterial blood gas analysis findings, baseline medication, and 6-minute walk test were recorded.

Operation related parameters (duration of operation, duration of cardiopulmonary bypass and bleeding volume) were recorded. Postoperative adverse events such as duration of ICU stay, postoperative duration of mechanical ventilation, pacemaker use, complicated infection and reintubations were recorded.

A full-night polysomnography as well as LG and related parameters were re-examined before discharge from hospital. The changes of AHIs, mean and lowest SPO2, LG and related parameters between pre- and post-operative polysomnography parameters were calculated.

The correlation between changes of polysomnography and LG parameters pre- and post-CPAP in CPAP group were analyzed. The correlation between changes of polysomnography and LG parameters pre- and post-operative in both CPAP and non-CPAP group were analyzed. The differences of polysomnography and LG parameters, and post-operative adverse events between CPAP and non-CPAP treatment group were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 years.
2. Patients with heart valve disease.
3. Patients combined with obstructive sleep apnea (apnea-hypopnea index >=5/h).
4. Received cardiac valve replacement surgery.
5. The enrolled patients having received patients' informed consent.

Exclusion Criteria:

1. History of stroke or clinical signs of peripheral or central nervous system disorders.
2. History of chronic obstructive pulmonary disease or asthma.
3. Enrolment in another clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
changes of apnea-hypopnea index | 14 days
  Changes of apnea-hypopnea index pre- and post-operative were compared between CPAP and non-CPAP patients.
changes of lowest SPO2 | 14 days
  Changes of lowest SPO2 pre- and post-operative were compared between CPAP and non-CPAP patients.
comparison of loop gain | 7 days
  Loop gain pre- and post-operative was compared between CPAP and non-CPAP patients.
  Loop gain pre- and post-CPAP treatment were compared in CPAP group.
arousal threshold | 14 days
  Arousal threshold pre- and post-operative was compared between CPAP and non-CPAP patients.
  Arousal threshold pre- and post-CPAP treatment were compared in CPAP group.
upper airway gain | 14 days
  Upper airway gain pre- and post-operative was compared between CPAP and non-CPAP patients.
  Upper airway gain pre- and post-CPAP treatment were compared in CPAP group.

SECONDARY OUTCOMES:
duration of operation | 12 hours
  Duration of operation was compared between CPAP and non-CPAP patients.
duration of cardiopulmonary bypass | 12 hours
  Duration of cardiopulmonary bypass was compared between CPAP and non-CPAP patients.
duration of ICU stays | 14 days
  Duration of ICU stays were compared between CPAP and non-CPAP patients.
duration of mechanical ventilation | 14 days
  Postoperative duration of mechanical ventilation was compared between CPAP and non-CPAP patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Wang, Ph D, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Ding N, Ni BQ, Zhang XL, Zha WJ, Hutchinson SZ, Lin W, Huang M, Zhang SJ, Wang H. Elimination of central sleep apnea by cardiac valve replacement: a continuous follow-up study in patients with rheumatic valvular heart disease. Sleep Med. 2014 Aug;15(8):880-6. doi: 10.1016/j.sleep.2014.02.007. Epub 2014 May 17. PMID 24938583
- [Background] Ding N, Ni BQ, Wang H, Ding WX, Xue R, Lin W, Kai Z, Zhang SJ, Zhang XL. Obstructive Sleep Apnea Increases the Perioperative Risk of Cardiac Valve Replacement Surgery: A Prospective Single-Center Study. J Clin Sleep Med. 2016 Oct 15;12(10):1331-1337. doi: 10.5664/jcsm.6182. PMID 27448416